CLINICAL TRIAL: NCT06541964
Title: The Effects of Parent-Provide Distraction and Windmill Toy Blowing Methods on Pain During Venous Blood Collection in Children Aged 6-12 Years
Brief Title: Two Different Distraction Methods for Reducing Procedural Pain in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Zeynep Erkut, Assistant Professor, PhD, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024/12-05
Record Dates: First submitted 2024-08-03; First posted 2024-08-07 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Procedural Pain
Keywords: Pain; Venous Blood Collection; Distraction
MeSH Terms: conditions — Pain, Procedural; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Parent-Provide Distraction Group (Experimental): Parent-Provide Distraction Group
  Interventions: Other: Parent-Provide Distraction
- Windmill Toy Blowing Group (Experimental): Windmill Toy Blowing Group
  Interventions: Other: Windmill Toy Blowing
- Control Group (Other): Control Group
  Interventions: Other: Control

INTERVENTIONS:
Other: Parent-Provide Distraction — The children will be asked riddles by their parents for 5 seconds before and during the blood collection procedure.
  Arms: Parent-Provide Distraction Group
Other: Windmill Toy Blowing — The children will blow on the windmill toy for 5 seconds before and during the blood collection procedure.
  Arms: Windmill Toy Blowing Group
Other: Control — No intervention will make on the children.
  Arms: Control Group

SUMMARY:
This research will be carried out in a randomized controlled experimental design in order to study the effect of parent-provide distraction and windmill toy blowing methods in reducing the pain caused by blood collection in children aged 6-12 who have applied to the children's blood collection unit. It will be taken by randomization so that there is no bias in the people who will be included in the study. Randomization table "https://www.calculatorsoup.com " it was created using.

After randomization, the children in the parent-provide distraction group with parental participation will be asked riddles by the parent during the venous blood collection procedure. The children in the windmill toy blowing group will blow a windmill toy during the venous blood collection process. For the children in the control group, no distraction will be made during venous blood collection. As soon as the procedure is completed, the pain score during the procedure and the pain score will be evaluated one minute after the procedure. The evaluation will be made by the child, parent and nurse who draws blood.

DETAILED DESCRIPTION:
Many different non-pharmacological methods are used to cope with adverse conditions such as pain caused by invasive procedures in children. One of these non-pharmacological methods is distraction. The American Pain Association recommends the use of distractions for pain control in children. By focusing the child's attention in another direction, the child's pain is controlled and reduced. As distraction methods, video games, virtual reality glasses, listening to music, watching cartoons, blowing balloons, reading books, blowing windmill toys, parent-provide distraction are used.

The aim of this study is to determine the effects of parent-provide distraction and windmill toy blowing in reducing pain during blood collection in children aged 6-12 years. Power analysis was performed to determine the number of people to be included in the research. The strength of the test was calculated using the G*Power 3.1 program. As a similar research in the relevant literature, the effect size of the difference in pain was calculated as 1.557 in the research conducted by Orhan (2020). In order to exceed the 95% value in determining the strength of the study, 51 people, including 17 people in groups with a significance level of 5% and an effect size of 1,557, must be reached (df=32; t=2,036). In the research, it was aimed to reach a total of 66 people, including 22 people in groups, taking into account the high strength of the test and the losses.

The Information Form, Wong Baker Faces Scale, VAS will be used for data collection. First of all, those who meet the criteria for inclusion in the research and research the purpose of the research will explain to the parents who volunteered to participate and their children by explaining the purpose of the research information about the research will be provided by the executor. Then about their participation in the study written and oral consent will be obtained from parents, and oral consent will be obtained from children. By obtaining information from the parent the information form will be filled out by the researcher before the blood collection procedure. Blood collection procedure it will be performed by a single experienced nurse Parental participation in the group of diverting attention information about the riddles will be provided by the researcher. By the research manager parents and children will be given information about the Wong Baker Faces Scale. Research manager children in the windmill toy blowing group will be supervised by blowing the windmill. No intervention will perform to reduce pain in the control group. In all groups, as soon as the procedure is completed and 1 minute after the procedure, the child's pain will be evaluated with the Wong Baker Faces Scale. The nurse and the parent will evaluate the child's pain with VAS. During the evaluation, pain assessments will be made in such a way that the child, parent and nurse will not see each other in order not to be affected by each other. It is estimated that the data collection process will take about 10-15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* The children whose between 6 and 12 years old,
* The children does not have a visual, hearing or mental problem,
* The children and the parent's knowledge of Turkish at the level of the mother tongue,
* The voluntary consent of the children and his/her parent to participate in the research.

Exclusion Criteria:

* The children whose younger than 6 years and older than 12 years,
* The children have a visual, hearing or mental problem,
* The children and the parent's inability to speak Turkish at the level of their native language,
* The children and the parent do not agree to participate in the research.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-11-13 (Actual)

PRIMARY OUTCOMES:
Pain Evaluated by Children (Wong-Baker Faces Scale) | During venipuncture procedure (when needle insertion and the first blood was seen in injector, until needle removed), and one minute after venipuncture procedure (one minute after the injector was removed)
  Pain will be assessed by children with Wong-Baker Faces Scale. It is a valid and safe individual notification-based scale used to describe pain in children aged 3-18 (Wong-Baker Faces Foundation-http://wongbakerfaces.org/). It consists of 6 facial expressions ranging from smiling face to crying facial expression, which are scored Dec Decently from 0 to 10 to describe the severity of pain. As the score obtained from the scale increases, the severity of pain increases, and the severity decreases as the score decreases. "Face 0" means that there is no pain. He has a smiley face expression. "Face 2" has a little pain. "Face 4 " has a little more pain. There are more than "face 6" pain. The "face 8" pain is quite a lot. The pain of "face 10" is unbearable. The severity of the pain can be defined by enabling children to choose the shape of the face from the expression of their pain.

SECONDARY OUTCOMES:
Pain Evaluated by Parents and Nurse (Visual Analog Scale) | During venipuncture procedure (when needle insertion and the first blood was seen in injector, until needle removed), and one minute after venipuncture procedure (one minute after the injector was removed)
  Pain will be assessed by parents and nurse with Visual Analog Scale. The scale developed by Freyd was used to determine the severity of pain. VAS is the scaled version of a 10-centimeter line from 1 to 10. a value of 10 indicates maximum pain, while a value of 0 means that there is no pain at all. He is asked to mark the appropriate place on the scale according to the level of pain. The pain score is determined by measuring with a ruler. This scale is a safe and widely used measurement tool accepted in the literature.

CONTACTS AND LOCATIONS:
Locations (1):
- Maltepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No